CLINICAL TRIAL: NCT07059715
Title: Mic Mac Study: A Prospective Study of Hemodynamic Coherence in Vasoplegic Syndrome After Cardiopulmonary Bypass
Brief Title: Mic Mac: Micro- and Macrocirculatory Assessment During Cardiac Surgery in Patients at Risk of Vasoplegic Syndrome: A Prospective Study.
Acronym: MicMac
Status: Recruiting | Type: Observational
Sponsor: European Georges Pompidou Hospital (Other)
Responsible Party: Principal Investigator, NOUGUE Hélène, Investigator Coordinator, European Georges Pompidou Hospital
Other Study IDs: 2024-A01235-42
Record Dates: First submitted 2025-02-21; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Vasoplegic Syndrome of Cardiac Surgery
Keywords: vasoplegia syndrome; post cardiopulmonary bypass; cardiac surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients at risk of vasoplegia syndrome after cardiac surgery: All patients at high risk of vasoplegia syndrome after cardiac surgery because they have cardiopulmonary bypass during the surgery

SUMMARY:
This research focuses on understanding the vasoplegic syndrome after cardiac surgery under extracorporeal circulation and in the aftermath of your surgery in the ICU.

The investigators evaluate variations in a number of clinical and biological parameters during cardiac surgery and in the 48 hours following resuscitation. In addition to all the monitors investigators usually use to monitor vital parameters during this type of procedure, investigators use sensors placed on the skin at the earlobe and palm of the hand to assess the quality of blood circulating in the body.

The investigators would like to know if these observations help us to better understand the vasoplegic syndrome (persistent drop in blood pressure requiring the administration of medication to maintain normal blood pressure), a known but poorly understood complication following cardiac surgery under extracorporeal circulation. Extracorporeal circulation is the pump that keeps the blood circulating in your body when the heart is stopped while the surgeon works on the heart.

DETAILED DESCRIPTION:
In 2019, 45,236 cardiovascular surgical procedures were performed in France. Despite improved surgical and anesthetic management, cardiovascular surgery continues to be associated with a high mortality rate, with an estimated in-hospital death rate of 5.8%. One of the major complications associated with the patient's condition and the complexity of the surgery is post-extracorporeal circulation vasoplegia syndrome, the incidence of which is estimated at between 5 and 44%. It is associated with a high mortality rate of around 40%. This vasoplegia results in arterial hypotension and organ damage, culminating in multivisceral failure and death. This phenomenon remains poorly understood, as it is extremely complex and multifactorial (vasodilation by pathological nitric oxide production, role of neprilysin, depletion of endogenous catecholamines, alteration of the autonomic nervous system). At present, the only treatments available to manage vasoplegic syndrome are symptomatic. This vasoplegia is the consequence of alterations in microreactivity, leading to a loss of hemodynamic coherence between the macrocirculation and the microcirculation.

The aim of this work is to identify the metabolic pathways responsible for the alterations in vasoreactivity that lead to this loss of hemodynamic coherence, manifesting as hypotension at preserved cardiac output and complicating organ failure.

The investigators will select patients at risk of vasoplegic syndrome after extracorporeal circulation. A detailed assessment of their microcirculatory and macrocirculatory function, combined with blood and urine biomarker assays reflecting circulatory status at the time of sampling, will be carried out before the start of surgery, at the various key stages of cardiovascular surgery, then immediately post-operatively, at 12 hours, 24 hours, and 50 hours from the end of surgery. The monitoring of these parameters, whether or not associated with the appearance of a vasoplegic syndrome following extracorporeal circulation, will enable the investigators to better characterize the elements undergoing modification, and thus to better target the markers and metabolic pathways involved in vasoplegic syndrome, which in turn will enable the proposal of targeted curative or even preventive therapies.

ELIGIBILITY:
Inclusion Criteria:

Have at least 3 point of the following risk factors for post-body circulation vasoplegic syndrome:

* Acute or chronic heart failure with left ventricular ejection fraction< 40% (1 pt)
* Complex cardiac surgery ( 2 pts)
* Cardiovascular risk factors with a EuroSCORE> 4% (1 pt)
* Chronic Kidney Disease Stage 4
* Type 2 Diabetes Mellitus
* Pre-operative heparin treatment
* Hypothyroidism
* Anti-hypertensive treatments including an ACE inhibitor, an angiotensin II receptor antagonist, a beta-blocker or Sacubitril

Exclusion Criteria:

* Heart transplantation
* Pre-operative hemodynamic instability
* Pregnant women
* Age <18
* Pre-existing sepsis
* Extracorporeal circulation support
* Heartmate/Impella/Carmat patient
* Hypothalamo-hypophyseal pathologies
* Adrenal insufficiency
* Anuric patient
* Guardianship/ curatorship
* Lack of social security coverage
* Opposition to clinical research by patients or their families

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population is all patients with risk factors at post operative vasoplegia syndrome (3 points or more in "inclusion criteria") who will have a cardiac surgery in the Georges Pompidou European Hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in blood neprilysin activity. | From enrollment (preoperative) to 48 hours after cardiac surgery
  Change from baseline in plasma neprilysin enzymatic activity measure at multiple timepoints with fluorimetry.
  Unit of Measure: pmol/mL/min
Change in blood neprilysin concentration | From enrollment (preoperative) to 48 hours after cardiac surgery
  Change from baseline in plasma neprilysin concentration measured at multiple timepoints with mass spectrometry.
  Unit of Measure: µg/L

SECONDARY OUTCOMES:
Change in cardiac output. | From enrollment (preoperative) to 48 hours after cardiac surgery.
  Change in cardiac output (L/min) assess using transthoracic, transesophageal ultrasound or invasive hemodynamic monitoring (FloTrac, Hemosphere,...).
Change in mean arterial pressure | From enrollment (preoperative) to 48 hours after cardiac surgery
  Mean arterial pressure is continuously monitor with an arterial catheter and record in mmHg.
Change un skin marbling score | From enrollment (preoperative) to 48 hours after cardiac surgery
  Marbling is assessed using a validated ordinal scale (from 0: no marbling to 5: intense marbling) on the anterior knee surface. Score changes is used to evaluate peripheral perfusion and microcirculatory system.
Change in skin recoloration time. | From enrollment (preoperative) to 48 hours after cardiac surgery
  Skin recoloration time is measured in seconds after fingertip pressure and a return to the initial skin color. This time reflects peripheral perfusion and microcirculatory status.
vasopressor requirement variation | From enrollment (preoperative) to 48 hours after cardiac surgery
  The dose of vasopressors (e.g: norepinephrine) administered is calculated in µg/kg/min, normalized to body weight and duration, to quantify circulatory support needs.
Change in tissue oxygen saturation. | From enrollment (preoperative) to 48 hours after cardiac surgery
  Tissue oxygen saturation (StO₂) is measured non-invasively on the forehead using near-infrared spectroscopy (NIRS) technology and reported in percentage (%).
Change in transcutaneous tissue CO₂ pressure | From enrollment (preoperative) to 48 hours after cardiac surgery
  Transcutaneous carbon dioxide (PtCO₂) is measured in mmHg using an earlobe sensor maintained at 37°C. This reflects local tissue perfusion and CO₂ clearance.
Change in plasma lactate concentration. | From enrollment (preoperative) to 48 hours after cardiac surgery
  Plasma lactate levels are measured in mmol/L from arterial blood samples. Lactate serves as a biomarker of tissue hypoperfusion and anaerobic metabolism.
Change in central venous oxygen saturation | From enrollment (preoperative) to 48 hours after cardiac surgery
  Mixed venous oxygen saturation (SvO₂) is obtained with central veinous blood samples. ScvO₂ is used to detect tissue hypoperfusion. Measure in percentage (%).
Change in venous-to-arterial CO₂ gap | From enrollment (preoperative) to 48 hours after cardiac surgery
  The central venous-to-arterial CO₂ gradient is calculated in mmHg by subtracting arterial from venous pCO₂, as an indicator of tissue perfusion.
Change in plasma creatinine level | From enrollment (preoperative) to 48 hours after cardiac surgery
  Plasma creatinine concentration was measured in µmol/L using standard enzymatic assays to assess renal function.
Change in B-type natriuretic peptide 1-32 | From enrollment (preoperative) to 48 hours after cardiac surgery
  BNP 1-32 concentrations were measured in pmol/L from plasma samples using mass spectrometry technique to assess cardiac strain.
Change in B-type natriuretic peptide | From enrollment (preoperative) to 48 hours after cardiac surgery
  Plasma B-type natriuretic peptide concentration was measured in ng/L using standard enzymatic assays to assess cardiac strain.
Change in NT-proBNP concentration | From enrollment (preoperative) to 48 hours after cardiac surgery
  NT-proBNP levels are measured in ngl/L from plasma samples using standard enzymatic assays as a marker of cardiac dysfunction.
Change in specific NT-proBNP 1-76 concentration | From enrollment (preoperative) to 48 hours after cardiac surgery
  NT-proBNP 1-76 fragment levels are measured in pmol/L from plasma samples using mass spectrometry as a marker of cardiac dysfunction.
Change in T71-glycosylated proBNP | From enrollment (preoperative) to 48 hours after cardiac surgery
  The percentage of T71-glycosylated proBNP is determined from plasma samples using mass spectrometry, representing the ratio of glycosylated to total proBNP forms.
Change in vasopressin level | From enrollment (preoperative) to 48 hours after cardiac surgery
  Plasma vasopressin levels are measured in pmol/L by immunoradiology to assess endogenous vasopressor response to circulatory stress.
Change in aldosterone level. | From enrollment (preoperative) to 48 hours after cardiac surgery.
  Plasma aldosterone concentrations are measured in pmol/L using immunoradiology to evaluate the activation of the renin-angiotensin-aldosterone system.
Change in angiotensin II level | From enrollment (preoperative) to 48 hours after cardiac surgery
  Plasma angiotensin II levels are quantified in pmol/L using mass spectrometry techniques to monitor vasoconstrictive hormonal activity and the activation of the renin-angiotensin-aldosterone system.
Change in endocan level | From enrollment (preoperative) to 48 hours after cardiac surgery
  Plasma endocan concentrations are measured in pmol/L with ELISA techniques to reflect endothelial activation and inflammation in kidney and lung.
Change in 5-MTP level. | From enrollment (preoperative) to 48 hours after cardiac surgery
  Plasma 5-MTP levels were measured in nmol/L using high-performance liquid chromatography to evaluate to evaluate systemic metabolic stress.

CONTACTS AND LOCATIONS:
Overall Officials: Helene NOUGUE, MCUPH, Principal Investigator — Georges Pompidou European Hospital
Locations (1):
- Georges Pompidou European Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: . Gökdemir, Begüm Nemika, et Nedim Çekmen. " Vasoplegic Syndrome and Anaesthesia: A Narrative Review ". Turkish Journal of Anaesthesiology and Reanimation 51, no 4 (1 august 2023): 280 89. — https://doi.org/10.4274/TJAR.2023.221093
- See also: . Vodovar, Nicolas, Marie-France Séronde, Said Laribi, Etienne Gayat, Johan Lassus, James L. Januzzi, Riadh Boukef, et al. " Elevated Plasma B-Type Natriuretic Peptide Concentrations Directly Inhibit Circulating Neprilysin Activity in Heart Failure ". JA — https://doi.org/10.1016/j.jchf.2015.03.011